CLINICAL TRIAL: NCT05347589
Title: Effects of Post Isometric Relaxation of Quadratus Lumborum With and Without Gluteus Maximus Activation on Pain, Disability and Pelvic Tilt Angle in Patients With Innominate Upslip Suprapubic Dysfunction
Brief Title: PIR of Quadratus Lumborum With and Without Gluteus Maximus Activation in Innominate Upslip Suprapubic Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0129 Uzair
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Innominate Upslip Suprapubic Dysfunction
Keywords: sacroiliac joint; suprapubic dysfunction; Muscle pain; Innominate upslip; pelvis
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post isometric relaxation of quadratus lumborum and gluteus Gluteus maximus activation exercises (Experimental)
  Interventions: Other: Post isometric relaxation of quadratus lumborum and gluteus Gluteus maximus activation exercises; Other: post isometric relaxation of the Quadratus lumborum
- post isometric relaxation of the Quadratus lumborum (Active Comparator)
  Interventions: Other: post isometric relaxation of the Quadratus lumborum

INTERVENTIONS:
Other: Post isometric relaxation of quadratus lumborum and gluteus Gluteus maximus activation exercises — Post Isometric Relaxation: The patient will be in a left recumbent position with his leg in a fully flexed position close to his chest and fixed by his left hand. The patient is asked to hold the treatment table with a right hand in an overhead position to support the body in applying the technique. The patient fully extended left will be taken away from the treatment table. At this point, the patient will be asked to press the leg down until the range where the patient feels discomfort to the point of torsion of Quadratus lumborum. This is the point that is the barrier range. Smaller than this range the patient will be asked to lift his left against the counterforce by the therapist and hold it for five to seven seconds which will be followed by five to seven seconds of relaxation. The technique will be repeated by five times in the pain-free range.
  Arms: Post isometric relaxation of quadratus lumborum and gluteus Gluteus maximus activation exercises
Other: post isometric relaxation of the Quadratus lumborum — Post Isometric Relaxation: The patient will be in a left recumbent position with his leg in a fully flexed position close to his chest and fixed by his left hand. The patient is asked to hold the treatment table with a right hand in an overhead position to support the body in applying the technique. The patient fully extended left will be taken away from the treatment table. At this point, the patient will be asked to press the leg down until the range where the patient feels discomfort to the point of torsion of Quadratus lumborum. This is the point that is the barrier range. Smaller than this range the patient will be asked to lift his left against the counterforce by the therapist and hold it for five to seven seconds which will be followed by five to seven seconds of relaxation. The technique will be repeated by five times in the pain-free range

SUMMARY:
The innominate up slip dysfunction is the most common in athletes and non-athletes, who present with low back pain and sacroiliac dysfunction. The main muscular structure that forms the force closure of the joint involves the bicep femoris and gluteus maximus that are involved in the stability of the of the pelvis through immense attachments through the Sacro-tuberous ligament. The objective of this study is to determine the effectiveness of Post Isometric Relaxation (PIR) of Quadratus lumborum with and without Gluteus maximus activation on pain, disability and pelvic tilt angle in patients with innominate upslip suprapubic dysfunction.

The study will be a randomized controlled trial involving 34 patients both males and females aged 20 to 40 years with history of unilateral pelvic pain not radiating to L5 or above, Positive finding of sitting flexion test, standing flexion tests, stork test and Positive active straight leg raise test will be randomly recruited by consecutive sampling technique. The subjects having ankylosing spondylitis, lumbar radiculopathy, spinal pathologies, or any lumbar fracture will be excluded. All the patients in the study will be randomly assigned into two groups where Group A will be given muscle energy technique of quadratus lumborum along with gluteus maximus activation and Group B will be a control group treated with muscle energy technique only. Both groups will be given buttock squeezing and drawing in maneuver as common treatment along with muscle energy technique. Each session will be repeated for 20 minutes thrice a week. The treatment duration will be 4 weeks. Outcomes will be measured at the first day and then at the end of the 4th week by numeric pain rating scale, modified Oswestry disability index and iHandy inclinometer application. .

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 to 40 years
2. Both males & females
3. History of unilateral pelvic pain not radiating to L5 or above
4. Positive finding of sitting flexion test, standing flexion tests, stork test.
5. Positive active straight leg raise test

Exclusion Criteria:

1. Subjects diagnosed with ankylosing spondylitis.
2. Lumbar radiculopathy
3. Spinal pathologies including spondylosis and spondylolisthesis.
4. Subjects immediately post pregnancy.
5. Disc herniation
6. Lumbar fractures or spinal surgeries

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-12-25 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4 weeks
  The numeric pain rating scale is a measurement of pain intensity in adults. The NPRS is a segmented numeric version of visual analogue scale (VAS) in which respondent select a whole number (0 to 10) that best reflects the intensity of pain. Scores range from 0 to 10
Modified Oswestry disability index (MODI) | 4 weeks
  The disability will be measured by using the modified Oswestry Disability Index in individuals with innominate up slip suprapubic dysfunction. This is an extremely important tool used to measure a patient's permanent functional disability. The total score ranges from 0 to 50, with each section having a total possible score of 5. The patient can be further subcategorized into five groups according to their total score: 0%-20% (minimal disability), 20%-41% (moderate disability), 41%-60% (severe disability), 61%-80% (crippled), and 81%-100% (bedridden). The modified Oswestry Disability Index has a minimum charge of 15.5%. This measure has been proven to have good validity for detecting changes in the SIJ, with a minimum difference of 13-15 indicating clinical significance
I-Handy level inclinometer mobile app | 4 weeks
  The iPhone 12 (Apple Inc, Cupertino, CA, USA) will be used as a measuring instrument with level application (iHandy level). The iHandy level application is integrated into the iPhone and is a free application with a visual display similar to that of a digital inclinometer in regard to numeric size. The application uses the iPhones built-in accelerometer and a digital display to display the angle measured.. The unit of measurement will be degrees

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Ghurki Trust Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Penalver UJ, Palop-Montoro MV, Manzano-Sanchez D. Effectiveness of the Muscle Energy Technique versus Osteopathic Manipulation in the Treatment of Sacroiliac Joint Dysfunction in Athletes. Int J Environ Res Public Health. 2020 Jun 22;17(12):4490. doi: 10.3390/ijerph17124490. PMID 32580480
- [Background] Sarkar M, Goyal M, Samuel AJ. Comparing the Effectiveness of the Muscle Energy Technique and Kinesiotaping in Mechanical Sacroiliac Joint Dysfunction: A Non-blinded, Two-Group, Pretest-Posttest Randomized Clinical Trial Protocol. Asian Spine J. 2021 Feb;15(1):54-63. doi: 10.31616/asj.2019.0300. Epub 2020 Jan 30. PMID 31992024
- [Background] Patel VD, Eapen C, Ceepee Z, Kamath R. Effect of muscle energy technique with and without strain-counterstrain technique in acute low back pain - A randomized clinical trial. Hong Kong Physiother J. 2018 Jun;38(1):41-51. doi: 10.1142/S1013702518500051. Epub 2018 Apr 4. PMID 30930578
- [Background] Kamali F, Zamanlou M, Ghanbari A, Alipour A, Bervis S. Comparison of manipulation and stabilization exercises in patients with sacroiliac joint dysfunction patients: A randomized clinical trial. J Bodyw Mov Ther. 2019 Jan;23(1):177-182. doi: 10.1016/j.jbmt.2018.01.014. Epub 2018 Jan 31. PMID 30691749
- [Background] Ghasemi C, Amiri A, Sarrafzadeh J, Dadgoo M, Jafari H. Comparative study of muscle energy technique, craniosacral therapy, and sensorimotor training effects on postural control in patients with nonspecific chronic low back pain. J Family Med Prim Care. 2020 Feb 28;9(2):978-984. doi: 10.4103/jfmpc.jfmpc_849_19. eCollection 2020 Feb. PMID 32318454
- [Background] Sanika V, Prem V, Karvannan H. Comparison of Glutues Maximus Activation to Flexion Bias Exercises Along with MET Technique in Subjects with Anterior Rotated Sacroiliac Joint Dysfunction-a Randomised Controlled Trial. Int J Ther Massage Bodywork. 2021 Mar 1;14(1):30-38. eCollection 2021 Mar. PMID 33654504
- [Background] Copay AG, Cher DJ. Is the Oswestry Disability Index a valid measure of response to sacroiliac joint treatment? Qual Life Res. 2016 Feb;25(2):283-292. doi: 10.1007/s11136-015-1095-3. Epub 2015 Aug 6. PMID 26245709
- [Background] Cana-Pino A, Espejo-Antunez L, Adsuar JC, Apolo-Arenas MD. Test-Retest Reliability of an iPhone(R) Inclinometer Application to Assess the Lumbar Joint Repositioning Error in Non-Specific Chronic Low Back Pain. Int J Environ Res Public Health. 2021 Mar 3;18(5):2489. doi: 10.3390/ijerph18052489. PMID 33802528